CLINICAL TRIAL: NCT05258162
Title: Comparison of Mobilization and Muscle Energy Technique in Patients With Post-Traumatic Elbow Stiffness
Brief Title: Comparison of Mobilization and MET Post-Traumatic Elbow Stiffness
Acronym: MET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah/RCRS/REC/00939
Record Dates: First submitted 2022-02-20; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Elbow Fracture
Keywords: Post Traumatic Elbow Stiffness; Pain; Elbow; Disability; Fracture
MeSH Terms: conditions — Elbow Fractures; Pain; Fractures, Bone | interventions — Range of Motion, Articular; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization (Experimental): Mobilizations are performed with minimum 6 seconds distraction stretch followed by partial release then followed by slow intermittent stretch at 3-4 seconds intervals.
  Oscillations for 2 minutes at 2-3 oscillations per second.
  Interventions: Other: Mobilization
- Muscle Energy Technique (Experimental): Muscle Energy Technique is given in the form of post isometric relaxation with 5-7 sec hold for 8-10 repetitions followed by a gentle passive stretch. Only 20% resistance is offered to the isometric contraction.
  Interventions: Other: Muscle Energy Technique

INTERVENTIONS:
Other: Mobilization — Hot pack for ten minutes.
  Active and active-assisted exercises for the:
  * Elbow flexion and extension
  * Wrist flexion and extension
  * Forearm supination and pronation
  * Lock and key exercises.
  * Shoulder flexion, extension, abduction, adduction, and rotation (10 repetitions x 1sets) Low-intensity isometric resistance exercises for;
  * Elbow flexion and extension
  * Forearm supination and pronation (10 sec hold) (10 repetitions x 1 set) Resistance will be provided manually by the therapist. Along all these exercises Mobilisations are performed with minimum 6 seconds distraction stretch followed by partial release then followed by slow intermittent stretch at 3-4 seconds intervals.
    3 days per week for 3 weeks. Oscillations for 2 minutes at 2-3 oscillations per second.
  Other Names: Hot pack; Range of Motion Exercises; Isometrics
  Arms: Mobilization
Other: Muscle Energy Technique — Hot pack for ten minutes.
  Active and active-assisted exercises for the:
  * Elbow flexion and extension
  * Wrist flexion and extension
  * Forearm supination and pronation
  * Lock and key exercises.
  * Shoulder flexion, extension, abduction, adduction, and rotation (10 repetitions x 1sets) Low-intensity isometric resistance exercises for;
  * Elbow flexion and extension
  * Forearm supination and pronation (10 sec hold) (10 repetitions x 1 set) Resistance will be provided manually by the therapist. Along all these exercises Muscle Energy Technique is given in the form of post isometric relaxation with 5-7 sec hold for 8-10 repetitions followed by a gentle passive stretch. Only 20% resistance is offered to the isometric contraction.
    3 days per week for 3 weeks.
  Other Names: Hot pack; Range of Motion Exercises; Isometrics
  Arms: Muscle Energy Technique

SUMMARY:
The purpose of this study is to find the effects of Mobilization and Muscle energy technique in patients with post-traumatic elbow stiffness.

DETAILED DESCRIPTION:
A randomized control trial was conducted at Benazir Bhutto Hospital, Rawalpindi. The sample size with reference to parent article was 10 calculated through open epi tool. But 30 patients were included in the study to increase the statistical power of analysis. The participants were divided into two interventional groups i.e. Group A and Group B, each having 15 participants. The study duration was 1 year. Sampling Technique applied was non probability purposive sampling technique. Random Allocation will be through sealed envelope method into two treatment group i.e. Group A and Group B. Only 18-35 years old patients (both male and female) with Post-traumatic elbow stiffness were included in the study. Tools that were used in the study are NPRS, DASH questionnaire, TAMPA scale and Goniometer. Total duration of treatment for both groups was 3 weeks, 3 days a week. Pre and post assessment was done. Data was analyzed through SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

* Patients with post-operative elbow stiffness after distal end extra-articular humerus fractures.
* Patients with proximal radius ulna fractures.
* Minimum immobilization period of 3 weeks

Exclusion Criteria:

* Any ligament injury
* Patients with Diabetes
* Patients with RA
* Patients with Pathological fractures
* Revision surgeries
* Neuro-vascular disorders.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 3rd week
  Changes from baseline Numeric pain rating scale is a self-administered, or analyst reported, measuring instrument comprising of a scale that shows numerical ranges usually from 0-10 or 0-100. In this scale extreme or farthest point shows having 'no pain' to having 'extreme pain'.
ROM Elbow (Flexion) | 3rd week
  Changes from baseline range of motion( ROM) of elbow joint flexion is taken by using Goniometer.
ROM Elbow (Extension) | 3rd week
  Changes from baseline range of motion( ROM) of elbow joint extension is taken by using Goniometer.
ROM Forearm (Supination) | 3rd week
  Changes from baseline range of motion( ROM) of forearm supination is taken by using Goniometer.
ROM Forearm (Pronation) | 3rd week
  Changes from baseline range of motion (ROM) of forearm pronation is taken by using Goniometer.

SECONDARY OUTCOMES:
Disability | 3rd week
  Changes from baseline disability is measured through DASH (Disability of the arm, shoulder and hand) questionnaire. DASH questionnaire is a self reported area specific outcome measuring tool for symptoms and disabilities in upper limb. It mainly comprise of a 30-items scale which is further consist of questions related to difficulty in performing normal daily activities, scored on 5 response options. Scores for these 30 items then calculate on a scale of 0 (no disability) to 100 (most severe disability)
kinesiophobia (fear of movement) | 3rd week
  Changes from baseline kinesiophobia is measured through Tampa scale which is a 17 item scale. Total scores of this scale ranges from 17-68. Where 17 means no kinesiophobia and 68 means severe kinesiophobia while score of ± 37 indicates that there is kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Benazir Bhutto Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No